CLINICAL TRIAL: NCT05027646
Title: A Randomized, Open-Label, Replicate Treatment, 2-Part, Crossover Study to Assess Bioequivalence and Adhesion Properties Between Two Granisetron Transdermal Patches Manufactured at Different Sites.
Brief Title: Study to Assess Bioequivalence and Adhesion Properties Between Two Granisetron Transdermal Patches.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 392MD/48/C
Record Dates: First submitted 2021-08-09; First posted 2021-08-30 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers
Keywords: Patch; Nausea; Anti-emetic; Granisetron
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, 2-part, open-label, crossover study in healthy subjects to establish BE (Part 1) and evaluate adhesion (Part 2) between granisetron transdermal patches.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 - Bioequivalence (Experimental): Bioequivalence will be measured in approximately 42 healthy male and female subjects at a single center in the US to achieve at least 33 completers.
  Interventions: Drug: Sancuso - Part 1
- Part 2 - Adhesion (Experimental): Adhesion will be measured in approximately 90 healthy male and female subjects are planned to be enrolled at a single center in the US.
  Interventions: Drug: Sancuso - Part 2

INTERVENTIONS:
Drug: Sancuso - Part 1 — Part 1 - A Potent anti-emetic and highly selective antagonist of 5-HT3 receptors.
  Other Names: Granisetron Transdermal Patch
  Arms: Part 1 - Bioequivalence
Drug: Sancuso - Part 2 — Part 2 - A Potent anti-emetic and highly selective antagonist of 5-HT3 receptors.
  Other Names: Granisetron Transdermal Patch
  Arms: Part 2 - Adhesion

SUMMARY:
The study is designed to evaluate the BE and adhesion properties of granisetron transdermal patches manufactured at 2 different sites. The study has been designed in accordance with the FDA Guidance for Industry. Bioequivalence will be based on the Cmax and AUC to determine the peak and total drug exposure, respectively.

DETAILED DESCRIPTION:
This is a single-center, randomized, 2-part, open-label, crossover study in healthy subjects to establish bioequivalence (Part 1) and evaluate adhesion (Part 2) between granisetron transdermal patches manufactured at 2 different sites (Sancuso [test] and Sancuso [reference]).

Each part of the study will consist of a screening period, check-in days, treatment periods, washout period (Part 1 only), and an end-of-study visit. The duration of subject participation, excluding screening, for Part 1 is approximately 39 days and for Part 2 is approximately 17 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 55 years, inclusive
* BMI 18 to 30 kg/m2
* Healthy volunteers, health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results and physical examination.
* Agrees to comply with all protocol requirements.
* Able to provide written and voluntary informed consent.
* Female participants of childbearing potential have a negative pregnancy test and agree to adhere to an acceptable methods of birth control.
* Male participants with female partners of childbearing potential agree to acceptable methods of birth control.

Exclusion Criteria:

Participant to be excluded if,

* Presents with baseline systolic blood pressure >140 mm Hg and diastolic blood pressure >90 mm Hg.
* Any clinically significant ECG finding or QTcF interval >450 msec for males and >470 msec for females.
* A history of sensitivity to granisetron or other components of the transdermal patch.
* Pregnant or breastfeeding.
* Severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results, as determined by the investigator.
* Participants with following pre-existing liver functioning test elevations will be excluded: alanine aminotransferase or aspartate aminotransferase elevation >2 × ULN, and/or bilirubin >2 × ULN
* Acute or chronic renal or hepatic impairment, that may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results, as determined by the investigator.
* Acute or chronic psychiatric condition, including, but not limited to compulsive-depressive disorders, anxiety, and/or sleep disorders that may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results.
* A history of coronary heart disease, arterial or pulmonary hypertension, supraventricular or ventricular tachycardias, or other arrhythmias or heart rhythm and conduction disorders.
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or HIV types 1 or 2 antibodies at screening.
* If used any prescription (excluding hormonal birth control) or over the counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before the first application of the transdermal patch.
* If used 5-HT3 receptor antagonists and other serotonergic drugs (eg, selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors, monoamine oxidase inhibitors, mirtazapine, fentanyl, lithium, tramadol, and IV methylene blue) within 14 days before the first application of the transdermal patch.
* If used antihistamines within 72 hours prior to patch application or systemic or topical corticosteroids within 3 weeks before the first application of the transdermal patch.
* Present with a dermatological disorder at any relevant patch application site that precludes proper placement or may interfere with adhesion, site assessment, or potentially affect drug absorption.
* Has allergies or other contraindications to transdermal systems or patch adhesives or to medical adhesive tape, adhesive dressings, or other skin patches.
* If not willing to allow hair to be removed or clipped at the proposed patch application sites that may prevent proper placement of the patch.
* If presents with and has oily skin or any skin problems such as being damaged (cut or scraped) or irritated (redness or a rash) at the application sites.
* If consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or alcohol-, caffeine-, or xanthine containing products within 48 hours before the first application
* The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 3 months before the first application of the transdermal patch.
* If has a history of alcohol abuse or drug addiction within a year.
* If presents with a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking).
* If involved in strenuous activity or contact sports within 24 hours before the first application and during the study.
* If donated blood or blood products >450 mL within 30 days before the first application.
* If has a history of relevant drug and/or food or significant food allergy that could preclude a standard diet in the CRU.
* If received study drug in another investigational study within 30 days of the first application.
* In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve AUC (0-t) | 6 months
  AUC from time 0 to the time of the last measurable plasma concentration, calculated using the linear trapezoidal rule
Area under the plasma concentration versus time curve AUC (0-inf) | 6 months
  AUC from time 0 extrapolated to infinity, calculated as (AUC 0-t + [Clast/λz]) where Clast is the last measurable plasma concentration
Peak Plasma Concentration (Cmax) | 6 months
  Maximum concentration after dosing
Maximum concentration (Tmax) | 6 months
  Time to reach the maximum plasma concentration after dosing (Tmax)
T1/2 | 6 months
  Terminal phase half-life
CL/F | 6 months
  Total clearance after dosing
Vz/F | 6 months
  Apparent volume of distribution during the terminal phase, calculated as (CL/F)λz
Mean adhesion score (FDA scale) | 6 months
  Adhesion of the patch to the skin is assessed by the FDA 0-4 scoring system. The scoring for adhesion is: 0 = ≥ 90% adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% adhered (less than half of the patch lifting off the skin), 3 = > 0% to < 50% adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely off the skin). Adhesion is assessed daily when patches are insitu. The mean adhesion score will be derived from its individual adhesion scores at each assessment time point, averaged across all the equally spaced time points (except baseline timepoint). Difference in mean adhesion score between test and reference transdermal patches will be compared using a mixed-model analysis of variance.

SECONDARY OUTCOMES:
Number of subjects with treatment related adverse events will be as assessed as mild, moderate or severe and will be summarized descriptively and presented as frequency and percentage. | 6 Months
  Actual values and changes from baseline for clinical laboratory test results, vital sign measurements and 12-lead ECG results will be summarized by test and reference patches at each time point using descriptive statistics (number of subjects, mean, SD, median, minimum and maximum)
Adhesion performance score (FDA Scale) | 6 Months
  Adhesion of the patch to the skin is assessed by the FDA 0-4 scoring system. The scoring for adhesion is: 0 = ≥ 90% adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% adhered (less than half of the patch lifting off the skin), 3 = > 0% to < 50% adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely off the skin). Adhesion is assessed daily when patches are insitu. Proportion of subjects with adhesion performance score of interest will be compared between the test and reference transdermal patches. Time to mean adhesion score more than or equal to 2 will be investigated graphically if data warrant.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Bioavailability and Bioequivalence Studies Submitted in NDAs or INDs - General Considerations (DHHS 2014). U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER). March 2014
- [Background] Guidance for Industry: Assessing Adhesion With Transdermal and Topical Delivery Systems for ANDAs (DHHS 2018). U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER) October 2018